CLINICAL TRIAL: NCT02384473
Title: Real-Time Contrast Enhanced Ultrasound and Ultrasound-Based Elastography: Novel Quantitative Imaging Techniques for Early Therapy Response Assessment in Sarcomas
Brief Title: Real-Time Contrast-Enhanced Ultrasonography and Shear Wave Elastography in Predicting Treatment Response in Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11S-14-1; NCI-2014-02579 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00792; 11S-14-1 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-03-10 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Adult Soft Tissue Sarcoma; Bone Sarcoma; Retroperitoneal Sarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Real-time CEUS and SWE (Experimental): Patients undergo real-time CEUS and SWE at baseline, 6 weeks after initiation of neoadjuvant therapy, and 9 weeks after initiation of neoadjuvant therapy (prior to surgery).
  Interventions: Procedure: Real-Time CEUS; Procedure: SWE; Drug: Definity Suspension for Injection; Device: Philips Shear Wave Elastography

INTERVENTIONS:
Procedure: Real-Time CEUS — Undergo real-time CEUS
Procedure: SWE — Undergo SWE
  Other Names: Shear Wave Elastography
Drug: Definity Suspension for Injection — Participant will receive contrast agent by intravenous administration
  Other Names: Perflutren Lipid Microsphere
Device: Philips Shear Wave Elastography — Type of equipment used for SWE
  Other Names: Shear Wave Elagstography

SUMMARY:
This pilot clinical trial studies real-time contrast-enhanced ultrasonography and shear wave elastography in predicting treatment response in patients with soft tissue sarcomas. Ultrasonography and elastography are diagnostic imaging tests that use sound waves to make pictures of the body without using radiation (x-rays). Real-time contrast-enhanced ultrasonography and shear wave elastography may help measure a patient's response to treatment given before surgery in patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate whether two different radiologists can reliably interpret the following quantitative criteria regarding the maximally enhancing portion of a soft tissue sarcoma (STS), on sequential contrast-enhanced ultrasound (CEUS) exams performed before, during, and after neoadjuvant chemotherapy (NAC): change in peak enhancement (decibels), change in slope of enhancement curve, and change in area under the curve.

II. To evaluate CEUS as a potential early response assessment biomarker by comparing the CEUS rating result to computed tomography (CT)/magnetic resonance imaging (MRI) rating results. (Exploratory) III. To examine the agreement between CEUS versus CT/MRI determined treatment response within each radiologist rater. (Exploratory) IV. To examine the agreement between CEUS versus CT/MRI determined treatment response based on the consensus rating result from the two radiologist raters. (Exploratory) V. To explore potential quantitative biomarker from all possible parameters that can be extracted from CEUS data for assessing an early treatment response to neoadjuvant therapy (NAT) in sarcoma using receiver operating characteristic (ROC) curve when predicting radiologists rated binary outcome: responders versus non-responders. (Exploratory) VI. To collect preliminary data for shear wave elastography (SWE) in the same patient population. (Exploratory)

OUTLINE:

Patients undergo real-time CEUS and SWE at baseline, 6 weeks after initiation of neoadjuvant therapy, and 9 weeks after initiation of neoadjuvant therapy (prior to surgery).

After completion of study, patients are followed up at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy and/or conventional imaging (CT/MRI) proven STS or bone sarcoma with a measurable soft tissue component; these include patients with extremity, retroperitoneal, chest wall, or head and neck primary sarcomas
* Patients who are potential candidates to receive neoadjuvant therapy with either chemotherapy alone, radiation alone, immunotherapy alone or combined treatment with any of these modalities. If on therapy, patients in whom a new treatment protocol or modality is being considered.
* Patients competent to sign study specific informed consent
* Patients willing to comply with protocol requirements

Exclusion Criteria:

* Patients who are pregnant
* Patients who have a known cardiac shunt or pulmonary hypertension
* Patients with any known hypersensitivity to perflutren agent
* Patients who cannot consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Inter-reader agreement for sequential contrast-enhanced ultra sound for evaluating treatment response as determined by kappa coefficient | Up to 9 weeks
  Kappa coefficient will be used. Reviewer 1 will first rate the treatment response followed by reviewer 2. Reviewer 2 will be blinded to the rating of reviewer 1.

CONTACTS AND LOCATIONS:
Overall Officials: Mittul Gulati, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States